CLINICAL TRIAL: NCT01408862
Title: Effects of Incretins on Human Platelet Function
Status: Completed | Type: Observational
Sponsor: National Council of Scientific and Technical Research, Argentina (Other Government)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Carlos Jose Pirola, Investigador Superior, Director, National Council of Scientific and Technical Research, Argentina
Other Study IDs: INC-PL-01
Record Dates: First submitted 2011-08-01; First posted 2011-08-03 (Estimated); Results first posted 2014-09-23 (Estimated); Last update posted 2014-09-23 (Estimated); Status verified 2014-09

CONDITIONS: Inhibition of Platelet Aggregation by Incretins
Keywords: GLP1; GIP; platelets; human; aggregation

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- controls: Healthy volunteers will be asked to donor a 10-80 ml blood through a venous puncture
  Interventions: Other: venous puncture

INTERVENTIONS:
Other: venous puncture — Blood for in vitro studies will be drawn
  Other Names: volunteers

SUMMARY:
Novel drugs for the treatment of patients with diabetes are of interest for cardiologists if they reduce the risk of cardiovascular events. However, as documented by the current discussion about the potential benefits of glitazones, high hopes can fail. Initial beneficial cardiovascular effects shown in proof-of-concept studies were muted by the apparent higher mortality in the metaanalysis of studies with rosiglitazone. The rapidly increasing use of GLP-1 analogues and DPP-4 (Dipeptidyl protease 4) inhibitors for the treatment of type 2 diabetes mellitus may be of major interest for the cardiologist. Potential beneficial actions on the cardiovascular system so far shown in animal experiments and small proof of concept studies may provide the rationale for using these drugs specifically in diabetic patients with secondary complications such as macrovascular disease or diabetic cardiomyopathy. Theoretically, these new therapies could also proof beneficial in patients with heart failure, independently of concomitant diabetes mellitus. However, many unanswered questions need to be addressed in the near future to extend the experimental findings to potential benefits of real life patients. In summary a new class of antidiabetic drugs, which could possibly directly influence cardiovascular effects of diabetes mellitus and thus possibly treat or even prevent life threatening complications has become available.

Then our working hypothesis was that incretins may have desirable cardiovascular outcomes through modulating platelet function. In order to test this hypothesis we propose to assess the presence of their specific receptors in isolated human platelets. In addition, we proposed to sudy the effect of the endogenous incretins (glucagon-like peptide 1 and gastric inhibitory peptide) on human platelet function isolated in a test tube.

DETAILED DESCRIPTION:
Aims and Methods: The prevalence of Type 2 diabetes (T2D) continues to increase globally and brings with it a parallel increase in the associated cardiovascular disease complications. Correction of platelet hyperactivity holds promise for this high-risk population of T2D patients by contributing to restore normal hemostasis, which has lead to the search for new antiagregant drugs. Then, our aim was to study whether incretins may modulate platelet function; for this purpose platelets from healthy subjects who were not taken any medication were studied. Besides, normal mature megakaryocytes obtained by culture of human cord blood derived-CD34+ hematopoietic progenitor cells were also studied.

For platelet function studies, platelet aggregation was tested in the absence and presence of different concentrations (10-9 M to 10-5 M) of glucagon-like peptide-1,GLP1-(7-36)NH2, and glucose-dependent insulinotropic polypeptide (GIP) agonist by a turbidimetricassay. The effect of 300 mg/dLglucose added to the media was also evaluated. GLP1R (glucagon-like peptide 1 receptor) and GIPR (GIP receptor) mRNA expression was evaluated by Real Time PCR in platelet and megakaryocyte total mRNA. The putative presence of their proteins was assayed by western blot and flow cytometry in both samples.

ELIGIBILITY:
Inclusion Criteria:

* Healthy blood donors

Exclusion Criteria:

* Diabetes
* Hypertension
* Morbid obesity
* Cardiovascular disease
* Hematological diseases and hyperlipidemia

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2012-12; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos J Pirola, PhD, Principal Investigator — Unidad Ejecutora IDIM-CONICET

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Platelets from 20 healthy human subjects who were not taken any medication in the previous 10 days were studied during 18 month in our institution.
Groups:
- Controls: 20 healthy volunteers were asked to donor a 10-80 ml blood through a venous puncture
  venous puncture: Blood for in vitro studies were drawn
Period: Overall Study
Arm/Group | Controls
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Platelets from healthy human subjects who were not taken any medication in the previous 10 days were studied. They were subjects with no characteristics of the Metabolic Syndrome components.
Groups:
- Controls: Platelets from healthy human subjects who were not taken any medication in the previous 10 days were studied. Blood samples (30 ml) were drawn with i) ACD-C (9:1, v/v) (7 mmol/L citric acid, 93 mmol/L citrate, 139 mmol/L dextrose, pH 6.4) for gene expression and western blot studies; ii) with 1% EDTA for flow cytometry and iii) with 3.8% sodium citrate for functional studies. Blood samples were centrifuged at 150 g for 10 min to obtain platelet-rich plasma (PRP).
Arm/Group | Controls
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (10)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Region of Enrollment [Number; unit: participants] — Ciudad Autonoma de Buenos Aires, Argentina
  participants
    Argentina | 20

OUTCOME MEASURES:

1. Primary Outcome: Expression of Glucagon Like Peptide -1 (GLP-1) and Gastric Inhibitory Peptide (GIP) Receptors in Normal Human Platelets
Description: 1.1 Measurement of GLP-1 and GIP receptors at the platelet RNA level by Real Time-PCR 1.2 GLP-1 and GIP receptors detection at the protein level: 1.2.1 Expression on platelet membrane by flow cytometry. 1.2.2 Detection in total platelet proteins by western-blot. Data of flow cytometry are provided below
Time Frame: Platelets drawn from a volunteer were evaluated 1 time (in 1-2 days)
Measure: Mean (Standard Deviation); unit: percentage of positive cells
Groups:
- Controls: Flow cytometry studies In order to test the presence of GLP1 and GIP receptors on normal platelet membrane, indirect immunodetection was carried out in platelet samples from 20 normal donors.
Arm/Group | Controls
Number analyzed (Participants) | 20
percentage of positive cells
  GLP1R | 3.73 (2.43)
  GIPR | 4.42 (1.70)
Statistical Analysis 1: Comparison: Controls; Results will be expressed as mean + SD from independent experiments. Statistical significance between means were determined by Wilcoxon-paired test. Variable will be log-transformed if they were not normally distributed. . We used the CSS/ Statistica program package, StatSoft V 6.0. This analysis applies to both GLP1R and GIPR categories; Test type: Superiority or Other; p = 0.04, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0

2. Primary Outcome: Changes in Basal or Aggregant-induced Platelet Activation (With and Without Glucose Added to the Media, 200 mg/dl, 400 mg/dL) by GLP-1-(7-36)NH2 and Its Metabolite (GLP-1-(9-36)NH2)and a GIP Agonist at Different Concentrations.
Description: 1 Direct effect of GLP-1-(7-36)NH2 and its metabolite (GLP-1-(9-36)NH2) and GIP agonist on platelet aggregation, with and without preincubation at different glucose concentrations.
  2. GLP-1-(7-36)NH2 and its metabolite (GLP-1-(9-36)NH2) and GIP agonist modulation (with and without 300 mg/dL glucose added to the media) of platelet activation and aggregation induced by classical platelet agonists such as ADP, collagen and bovine von Willebrand factor.
  Data points from various conditions were combined (averaged),
Time Frame: Platelets drawn from a volunteer will be evaluated 1 time (in 1-2 days)
Population: We assume that with 10 samples per condition divided in 5 categories (1 control plus 4 concentrations of GLP1 and GIP agonists) for a standardized difference of 0.5 between groups and a p=0.05, the statistical power would be higher than 90%. We used a similar design to test the effect of GLP1 and GIP agonists on platelet aggregants.
Measure: Mean (Standard Deviation); unit: % of Inhibition
Groups:
- Controls: Healthy volunteers were asked to donor a 10-80 ml blood through a venous puncture
  venous puncture: Blood for in vitro studies were drawn
Arm/Group | Controls
Number analyzed (Participants) | 20
% of Inhibition
  GLP1 | 0 (10)
  GIP | 0 (8)
Statistical Analysis 1: Comparison: Controls; Results will be expressed as mean + SD from independent experiments. Statistical significance between means were determined by two-way ANOVA with repeated measures on one factor, for variables measured in several consecutive times. Variable will be log-transformed if they were not normally distributed. Wilcoxon test for paired samples was used. The Statistica program package (StatSoft V 6.0) were used to perform these analyses, which applied to both GLP1R and GIPR agonist effect categories; Test type: Superiority or Other; p = 0.20, ANOVA; Mean Difference (Final Values) = 0

ADVERSE EVENTS:
Time Frame: 2 hours
Description: We pay attention to common minor complications of the venous puncture, such as small hematoma.
Arm/Group | Controls
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

LIMITATIONS AND CAVEATS:
Albeit at high concentrations presumably well above of the physiological range, the use of native and rapidly degradable forms of these peptides may impose a limitation of this study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less